CLINICAL TRIAL: NCT05814276
Title: San Rocco Study: an Observational Study on Implementation of the Non-pharmacological Therapies for People With Dementia Living in Nursing Home
Brief Title: San Rocco Study: Implementation of the Non-pharmacological Therapies for People With Dementia Living in Nursing Home
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Associazione Ginco Ticino (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 02
Record Dates: First submitted 2023-02-24; First posted 2023-04-14 (Actual); Last update posted 2023-04-14 (Actual); Status verified 2023-04

CONDITIONS: Nursing Home; Dementia; Staff
Keywords: nursing home staff; behavioral symptoms; burnout
MeSH Terms: conditions — Dementia; Behavioral Symptoms; Burnout, Psychological

STUDY DESIGN:
Intervention Model Description: Participants will attend ten sessions on the non-pharmacological therapies' methodology and implementation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- San Rocco group (Experimental): The San Rocco study encompasses a training on the non-pharmacological therapies' methodology.
  Interventions: Behavioral: Training on non-pharmacological therapies' methodology
- As usual control group (No Intervention): Participants will continue the usual care activities and non-pharmacological interventions already in use in the Nursing Homes without participating in the training.

INTERVENTIONS:
Behavioral: Training on non-pharmacological therapies' methodology — The San Rocco study encompasses a training on the non-pharmacological therapies' methodology. It allows the professional caregiver to methodological definition of the non-pharmacological interventions and a comparison of shared readings of the challenging behaviors by the group of colleagues. Participants will follow:
  * Five meetings, lasting 11 hours overall, on the multidimensional assessment, the shared readings of behavioral disorders of each person and identification of the objectives through the discussion of cases, and administration of non-pharmacological therapies within the framework of the personalization of the interventions
  * Five meetings, lasting five and a half hours, for the supervision of the staff which implement the non-pharmacological therapies.
  As usual control group Participants will continue the usual care activities and non-pharmacological interventions already in use in the Nursing Homes without participating in the training.
  Arms: San Rocco group

SUMMARY:
The goals of this clinical trial are 1) to estimate the number of professional caregivers and the time spent to carry out the non-pharmacological therapies for people with dementia and 2) to evaluate differences between professional caregivers trained and non-trained to non-pharmacological therapies for people with dementia in term of caregivers' burnout and well-being of people with dementia living in nursing home.

The main questions it aims to answer are:

* How long does it take professional caregivers to implement and carry out non-pharmacological therapies?
* How many caregivers are needed to start and carry out non-pharmacological therapies?
* Do the non-pharmacological therapies improve the quality of life of people with dementia?
* Do the non-pharmacological therapies reduce behavioral and psychological symptoms of dementia?
* Do the non-pharmacological therapies improve professional caregiver burnout, sense of competence and ethical climate in nursing home?
* Do the non-pharmacological therapies reduce family caregivers' stress?

Participants will attend ten sessions:

* five theoretical meetings on dementia and non-pharmacological therapies;
* five supervision meetings on the methodology for implementing non-pharmacological therapies based on discussions of cases.

The investigators will compare the experimental group with an usual care control group to see if there are improvements in term of the quality of life of the resident perceived by the team, professional caregivers burnout, sense of competence of the carers and the ethical climate at the workplace.

DETAILED DESCRIPTION:
The San Rocco study is a case-control study with two parallel arms aimed to estimate the number of professional caregivers and the time spent to carry out the non-pharmacological therapies for people with dementia and to evaluate the three- and six-months effectiveness of a training on non-pharmacological interventions, compared to usual care activities. Investigators have planned to involve two convenience samples. Experimental group: 18 professional caregivers and 18 people with dementia living in the San Rocco Special Care Unit for people with dementia (Canton of Ticino, Switzerland). Control group: 18 professional caregivers of the Nursing Homes attending the non-active group of the I-ACE study (ClinicalTrials.gov ID: NCT05710523).

The Nursing Homes' responsibles will verify the presence of the inclusion and exclusion criteria. This information will be promptly transferred and kept in an electronic archive protected by a password. Access to the personal computer containing the data will be protected by an access key.

ELIGIBILITY:
Inclusion Criteria:

* length of service more than six months

Exclusion Criteria:

* Presence of psychiatric illness or other medical condition that prevents participation in the training

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2022-02-11 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
Time to carry out non-pharmacological therapies | 240 days
  To estimate how much time (i.e., minutes per day) the professional caregivers take to carry out the non-pharmacological therapies for people with dementia.
Number of professional caregivers involved in non-pharmacological therapies | 240 days
  To estimate the number of professional caregivers required to carry out the non-pharmacological therapies for people with dementia.

SECONDARY OUTCOMES:
Professional caregivers' burnout | 180 days
  Change in professional caregivers' burnout, as measured by the Maslach Burnout Inventory (MBI), from baseline to first and second follow up. The investigators expect a significant difference in the experimental group compared with the control group. The Maslach Burnout Inventory is a self-administered questionnaire with scores ranging from zero to 132, with higher scores indicating more severe burnout symptoms.
Professional caregivers' sense of competence | 180 days
  Change in the professional caregivers' sense of competence, as measured by the Sense of Competence in Dementia Care Staff Scale (SCDS), from baseline to first and second follow up. The investigators expect a significant difference in the experimental group compared to the control group. The Sense of Competence in Dementia Care Staff Scale is a self-administered questionnaire with scores ranging from 17 to 68, with higher scores indicating higher self-perception of competence.
Quality of life of people with dementia | 180 days
  Change in the quality of life of people with dementia perceived from professional caregivers, as measured by the Quality of Life in Late-stage Dementia questionnaire (QUALID), from baseline to first and second follow up. The investigators expect a significant difference in the experimental group compared to the control group. The Quality of Life in Late-stage Dementia questionnaire is a self-administered questionnaire with scores ranging from 11 to 55, with higher scores indicating lower quality of life for people with dementia.
Professional caregivers' perception of social capital and ethical climate | 180 days
  Change in the professional caregivers' perception of social capital and ethical climate, as measured by the self-administered questionnaire Social capital and ethical climate at the Workplace of a hospital scale (SEW), from baseline to first and second follow up. The investigators expect a significant difference in the experimental group compared to the control group. The Social capital and ethical climate at the Workplace of a hospital scale is a self-administered questionnaire and it consists of three sub-scales: the higher the mean score of two sub-scales (social capital in the workplace and ethical leadership), the greater the participants' perceived favourable characteristics, and the higher the mean score of one sub-scale (exclusive workplace climate), the greater the participants' perceived unfavourable work environment characteristics.
Behavioral and psychological symptoms in dementia | 180 days
  Change in the behavioral and psychological symptoms in dementia (BPSD), as measured by the Neuropsychiatric Inventory Nursing Home (NPI-NH), from baseline to first and second follow up. TThe investigators expect a significant difference in the experimental group compared to the control group.The Neuropsychiatric Inventory Nursing Home was validated for interviewing the professional caregivers on twelve behavioural areas, including depression. The frequency [from one (rarely, less than once a week) to four (very often, once, or more per day)] and the severity [from one (mild) to three (severe)] of each BPSD are reported. The domain scores (frequency × severity) are added into the total score, ranging from zero to 144, with higher scores indicating more severe symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Rita Pezzati, Professor, Principal Investigator — Ginco Ticino Association
Locations (1):
- Fondazione Casa San Rocco, Morbio Inferiore, Switzerland